CLINICAL TRIAL: NCT05800444
Title: Single and Multiple Dose Escalation Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BAY 3283142 Given as Oral Tablets in Japanese Healthy Male Participants in a Randomized, Placebo-controlled, Single-blind, Group Comparison Design
Brief Title: A Study to Learn How Safe the Study Treatment BAY3283142 is, How it Affects the Body, How it Moves Into, Through and Out of the Body When Single and Multiple Amounts Are Taken as Tablets in Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 21938
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease; Healthy Volunteers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAY3283142 (low dose) (Experimental): Participants will receive BAY3283142 as single low dose on Day 1 followed by multiple doses for 7 days from Day 3 to Day 9.
  Interventions: Drug: BAY3283142
- BAY3283142 (medium dose) (Experimental): Participants will receive BAY3283142 as single medium dose on Day 1 followed by multiple doses for 7 days from Day 3 to Day 9 (optional arm).
  Interventions: Drug: BAY3283142
- BAY3283142 (high dose) (Experimental): Participants will receive BAY3283142 as single high dose on Day 1 followed by multiple doses for 7 days from Day 3 to Day 9.
  Interventions: Drug: BAY3283142
- Matching placebo (Placebo Comparator): Participants will receive a BAY3283142 matching placebo as single dose on Day 1 followed by multiple doses for 7 days from Day 3 to Day 9.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BAY3283142 — Oral administration as tablet.
  Arms: BAY3283142 (high dose); BAY3283142 (low dose); BAY3283142 (medium dose)
Other: Placebo — Oral administration as tablet.
  Arms: Matching placebo

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD).

The kidneys filter extra water and waste out of the blood and make urine. CKD is a long-term, progressive decrease in the kidneys' ability to work properly.

The study treatment BAY3283142 is under development for treating CKD. It works by activating a protein called soluble guanylate cyclase (sGC) that generates cGMP - a molecule that relaxes blood vessels and is thought to have beneficial effects in CKD.

The participants of this study will be healthy and will have no benefit from the intake of the study treatment. However, the study will provide information on how to use BAY3283142 in subsequent studies in people with CKD.

The main purpose of this study is to learn how safe the study treatment BAY3283142 is and how it affects the body in comparison to placebo when given as single and multiple amounts in healthy male participants in Japan. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

To do this, the study team will compare the number of participants who have medical problems after taking BAY3283142 with those participants who take placebo. These medical problems are called adverse events. The study doctors and their team keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

Another purpose of this study is to learn how the study treatment BAY3283142 moves into, through, and out of the body. To answer this, the study doctors and their team will take blood samples from the participants and measure:

* The average highest level of BAY3283142 in the blood (also called Cmax)
* The average total level of BAY3283142 in the blood (also called AUC).

Dependent on the treatment group, the participants will either take BAY3283142 or placebo as tablet once a day. A group of participants will start out by receiving a low amount of the study treatment. The study doctors will look at the results from these participants and then decide whether to increase the amount of the study treatment in the next group of participants. Researchers use dose escalation studies to learn about the safety of a specific amount before participants are given a higher amount.

Participants will be in the study for up to 7 weeks, including an in-house stay of up to 15 days. One test (screening) visit to the study center is planned before the start of treatment and one follow-up visit is planned after the end of treatment.

During the study, the study team will:

* check vital signs
* do physical examinations
* take blood and urine samples
* examine the participants' heart health using electrocardiogram (ECG)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 20 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12 lead ECG.
* Race: Japanese.
* body mass index (BMI) within the range 18.0 and 29.9 kg/m^2 (inclusive).
* Body weight equal or above 55 kg (inclusive).
* Male: Contraceptive use by men and female partners of male participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator.
* A history of clinically relevant diseases of any organs.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study interventions will not be normal.
* Participants with thyroid disorders as evidenced by assessment of thyroid stimulating hormone levels outside the normal reference range.
* Known hypersensitivity to the study interventions (active substances or excipients of the preparations, e.g., lactose).
* Known severe allergies (e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids), urticaria or significant non-allergic drug reactions.
* Relevant diseases within the last 4 weeks prior to the first intake of study intervention.
* Febrile illness within 2 weeks before the first intake of study intervention.
* Known tendency for vasovagal reactions (e.g., after venipuncture) or history of syncope.
* History of gastrointestinal surgery, with the exception of appendectomy (surgery at least 12 months before screening) and inguinal hernia repair (the surgery at least 12 months before screening with the documentation of no intestine necrosis and no intestine segment resection, and participants must be fully recovered and have no signs or symptoms).
* Acute diarrhea or constipation within 14 days before the first intake of study intervention.
* Regular use of medicines.
* Use of any other systemic or topical medicines or substances which oppose the study objectives.
* Regular use of therapeutic or recreational drugs, e.g., carnitine products, anabolics, high dose vitamins.
* Excluded therapies (e.g., physiotherapy, acupuncture, etc.) within 1 week before the first intake of study intervention.
* Participation in another clinical study of an investigational drug (last dose) within 90 days or 5 half lives of the investigational drug, whichever is longer, before the first dose of this study.
* Exclusion periods from other studies or simultaneous participation in other clinical studies.
* Previous treatment during this study (allowing previously treated participants to be re included into the study may lead to bias).
* Clinically relevant findings in the 12-lead ECG such as a second- or third-degree atrioventricular block, prolongation of the QRS complex over or equal to 120 msec, or of the QTcF or QTcB intervals over 450 msec.
* Clinically relevant arrhythmic disturbances as found in the 12-lead ECGs (especially repeated supra- and ventricular ectopic beats - Lown classification grade 2 or more); known congenital QT prolongation.
* Systolic blood pressure (SBP) below 100 or above 140 mmHg (after 15 min of supine rest).
* Diastolic blood pressure (DBP) below 50 or above 90 mmHg (after 15 min of supine rest).
* Heart rate (HR) below 45 or above 90 bpm (after 15 min of supine rest).
* Clinically relevant findings in the physical examination.
* Positive results for HBsAg, anti-HCV, HIV antigen and antibody, and syphilis (cardiolipin-lecithin antigen, Treponema pallidum antibody).
* Creatine kinase (CK) above upper limit of normal (ULN), except marginal explainable changes which are expected to normalize before study intervention intake.
* Lipase and amylase above ULN (except isolated marginal increases of lipase or amylase to account for variability of the parameters, and the participant is asymptomatic and has no other laboratory changes assuming disease based on medical judgment).
* Glycosylated hemoglobin (HbA1c), serum creatinine, C-reactive protein (CRP), liver enzymes (e.g., alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, gamma-glutamyl transferase, total bilirubin) above ULN.
* Deviations from normal ranges of any other safety laboratory parameter indicating apparent disease (or for which disease cannot be excluded) or impacting the objectives of the study.
* Positive urine drug screening indicating drug abuse.
* Positive alcohol breath test.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 7 days after end of treatment with study intervention, an average of 18 days

SECONDARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity (AUC) after single (first) dose of BAY3283142 on Day 1 | 0 to 48 hours post-dose
Maximum observed drug concentration (Cmax) after single (first) dose administration of BAY3283142 on Day 1 | 0 to 48 hours post-dose
AUC during any dose interval after (last) multiple doses of BAY3283142 on Day 9 (AUCτ,md) | 0 to 24 hours post-dose
  An interval of 24 h will be used for τ (Tau).
Maximum observed drug concentration in measured matrix after (last) multiple doses of BAY3283142 on Day 9 (Cmax,md) | 0 to 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.